CLINICAL TRIAL: NCT05295823
Title: Patient Self Measurement of Post-Void Residual Bladder Volume (PVR) Using Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Butterfly Network, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 2000031258
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Voiding Disorders; Voiding Dysfunction
Keywords: post void residual bladder volume; portable usltrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participant will be blinded to the results of the Urologic healthcare provider's measurements; and the Urologic healthcare provider will be blinded to the results of the patient's measurements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Healthcare provider performed standard PVR measurement using existing ultrasound technology (No Intervention): The Urologic healthcare provider will perform standard point-of-care PVR measurement on the participant (3 consecutive measurements during the same encounter) using existing ultrasound technology
- Healthcare provider performed PVR measurement using Butterfly and bladder ultrasound images (Experimental): The Urologic healthcare provider will perform PVR measurement on the participant (3 consecutive measurements during the same encounter) using the Butterfly and bladder ultrasound images
  Interventions: Device: Butterfly portable ultrasound device with bladder ultrasound images
- Healthcare provider performed PVR measurement using Butterfly and abstract bladder images (Experimental): The Urologic healthcare provider will perform PVR measurement on the participant (3 consecutive measurements during the same encounter) using the Butterfly and abstract bladder images
  Interventions: Device: Butterfly portable ultrasound device with abstract bladder images
- Self PVR measurement using Butterfly and bladder ultrasound images (Experimental): The participant will perform self PVR measurement (3 consecutive measurements during the same encounter) using the Butterfly and bladder ultrasound images (prior to catheterization, if needed)
  Interventions: Device: Butterfly portable ultrasound device with bladder ultrasound images
- Self PVR measurement using Butterfly and abstract bladder images (Experimental): The participant will perform self PVR measurement (3 consecutive measurements during the same encounter) using the Butterfly and abstract bladder images (prior to catheterization, if needed)
  Interventions: Device: Butterfly portable ultrasound device with abstract bladder images

INTERVENTIONS:
Device: Butterfly portable ultrasound device with bladder ultrasound images — Point-of-care PVR measurement using existing ultrasound technology (3 consecutive measurements during the same encounter) the Butterfly portable ultrasound device with bladder ultrasound images
  Arms: Healthcare provider performed PVR measurement using Butterfly and bladder ultrasound images; Self PVR measurement using Butterfly and bladder ultrasound images
Device: Butterfly portable ultrasound device with abstract bladder images — Point-of-care PVR measurement using the Butterfly portable ultrasound device with abstract bladder images
  Arms: Healthcare provider performed PVR measurement using Butterfly and abstract bladder images; Self PVR measurement using Butterfly and abstract bladder images

SUMMARY:
This study would be the first to demonstrate feasibility, accuracy, reliability, clinical care impact, and patient satisfaction with remote monitoring of post-void residual bladder volume (PVR) using the Butterfly portable ultrasound device in patients with obstructive voiding dysfunction.

DETAILED DESCRIPTION:
This study would be the first to demonstrate feasibility, accuracy, reliability, and patient satisfaction with self measurement of PVR using the Butterfly portable ultrasound device.

In the current study protocol, participants will undergo routine clinical care with no additional clinical encounters for the purposes of this study. As part of routine clinical care, the patient will undergo 3 sequential measurements of patient PVR by the Urologic healthcare provider using the existing ultrasound technology, and a possible bladder catheterization for actual bladder volume measurement and to drain the bladder. Note that 3 sequential measurements are taken from which a mean and standard deviation are derived due to operator and technology-related variability in bladder volume measurement using ultrasound. Participants in the study will also undergo 3 sequential measurements of patient PVR by the Urologic healthcare provider using the Butterfly portable ultrasound device with ultrasound images of the bladder, and 3 sequential measurements of patient PVR by the Urologic healthcare provider using the Butterfly portable ultrasound device with abstract images of the bladder; and the participant will take 3 sequential self-measurements of PVR using the Butterfly portable ultrasound device with ultrasound images of the bladder and 3 sequential self-measurements of PVR using the Butterfly portable ultrasound device with abstract images of the bladder during the same clinic encounter. The Urologic healthcare provider might also perform a bladder catheterization of the patient to determine the actual PVR and to drain the bladder of the residual urine.

Ultimately, successful remote measurement of patient PVR may lead to a paradigm shift in how patients with voiding dysfunction are clinically monitored; and would be a critical tool in triaging patients with possible urinary retention at any time but most especially during a pandemic necessitating social distancing and judicious allocation of healthcare resources. Remote PVR measurement in patients with obstructive voiding dysfunction may lead to more accurate monitoring for urinary retention; early detection of and intervention for urinary retention and potential prevention of sequelae such as urinary tract infection/urosepsis, renal failure, and bladder failure; potential reduction in medical costs and travel burden by reducing unnecessary clinic and emergency room visits as well as the costs of treating potential sequelae of urinary retention; and better quality of life for patients with obstructive voiding dysfunction.

Ultrasound technology is non-invasive, uses sound waves (non-ionizing radiation) to produce a volume measurement, and is an exceptionally safe method of imaging with a very limited risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Patient with capacity to consent to the study and completion of informed consent document
* Ability to speak and read English

Exclusion Criteria:

* Patient without capacity to consent to the study or incompletion of informed consent document
* Inability to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of self-measurement of PVR using the Butterfly with bladder ultrasound images compared to the Butterfly with abstract bladder images measured by Bland-Altman analysis. | up to 6 months
  Accuracy of the patient self-measurement of PVR using the Butterfly portable ultrasound device with bladder ultrasound images compared to the Butterfly portable ultrasound device with abstract bladder images during the same encounter. It is measured by Bland-Altman analysis which describes agreement between two quantitative measurements. More agreement means less difference between measurements.
Accuracy of self-measurement of PVR using the Butterfly with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the Butterfly with bladder ultrasound images measured by Bland-Altman analysis. | up to 6 months
  Accuracy of the patient self-measurement of PVR using the Butterfly portable ultrasound device with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the Butterfly portable ultrasound device with bladder ultrasound images during the same encounter. It is measured by Bland-Altman analysis which describes agreement between two quantitative measurements. More agreement means less difference between measurements.
Accuracy of self-measurement of PVR using the Butterfly with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the Butterfly with abstract bladder images measured by Bland-Altman analysis. | up to 6 months
  Accuracy of the patient self-measurement of PVR using the Butterfly portable ultrasound device with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the Butterfly portable ultrasound device with abstract bladder images during the same encounter. It is measured by Bland-Altman analysis which describes agreement between two quantitative measurements. More agreement means less difference between measurements.
Accuracy of patient self-measurement of PVR using the Butterfly with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the existing ultrasound technology measured by Bland-Altman analysis. | up to 6 months
  Accuracy of the patient self-measurement of PVR using the Butterfly portable ultrasound device with bladder ultrasound images compared to the healthcare provider's measurements of patient PVR using the existing ultrasound technology during the same encounter. It is measured by Bland-Altman analysis which describes agreement between two quantitative measurements. More agreement means less difference between measurements.
Accuracy of patient self-measurement of PVR using the Butterfly with bladder ultrasound images compared to the healthcare provider's bladder catheterization of the patient measured by Bland-Altman analysis. | up to 6 months
  Accuracy of the patient self-measurement of PVR using the Butterfly portable ultrasound device with bladder ultrasound images compared to the healthcare provider's measurements from bladder catheterization of the patient during the same encounter. It is measured by Bland-Altman analysis which describes agreement between two quantitative measurements. More agreement means less difference between measurements.

SECONDARY OUTCOMES:
Patient Reported Outcomes Questionnaire to asses ease of use, satisfaction, and preference of Butterfly Device | up to 6 months
  Patient Reported Outcomes Questionnaire to assess patient-reported ease of use, satisfaction, and preference between using bladder ultrasound images or abstract bladder images for self measurement of PVR with the Butterfly device using a patient questionnaire at the conclusion of patient self measurements. A mix of open-ended and multiple-choice questions using a 5-point Likert scale of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Cavallo, MD, MPHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No